CLINICAL TRIAL: NCT00043537
Title: Treatment of Childhood Social Phobia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Central Florida (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Deborah Beidel, Professor of Psychology, University of Central Florida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH053703 (NIH); R01MH053703 (NIH)
Record Dates: First submitted 2002-08-09; First posted 2002-08-12 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Social Phobia
Keywords: Phobic Disorders; Mutism
MeSH Terms: conditions — Phobia, Social; Phobic Disorders; Mutism | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Social Effectiveness Therapy for Children (Experimental): Social Effectiveness Therapy for Children includes social skills training, peer generalization experiences and exposure therapy
  Interventions: Behavioral: Social Effectiveness Therapy for Children (SET-C)
- Fluoxetine (Experimental): Fluoxetine given in 10mg doses, up to 40 mg as tolerated
  Interventions: Drug: Fluoxetine
- Pill placebo (Placebo Comparator): Capsules identical to fluoxetine given in "10 mg." doses up to 40 mg.
  Interventions: Drug: Pill Placebo

INTERVENTIONS:
Behavioral: Social Effectiveness Therapy for Children (SET-C)
  Arms: Social Effectiveness Therapy for Children
Drug: Fluoxetine
  Arms: Fluoxetine
Drug: Pill Placebo
  Arms: Pill placebo

SUMMARY:
This 4-year study will compare the long-term effectiveness of behavioral treatment, fluoxetine (Prozac®), and placebo for treatment of social phobia in children and adolescents.

DETAILED DESCRIPTION:
Social phobia affects 3-5 percent of children, and prevalence rises with age. Youth with social phobia fear many activities that are part of everyday life and suffer from problems such as headaches or stomachaches, panic, avoidance, general anxiety, depression, loneliness, and a very restricted range of social relationships. Recent findings indicate a new psychosocial treatment called Social Effectiveness Therapy for Children (SET-C) is effective in treating children ages 8-11, resulting in reduced emotional distress and improved social functioning. Treatment effects have been maintained for up to 6 months. This study will examine SET-C in children ages 8-15. Because available data suggest that the drug fluoxetine is a promising treatment, SET-C will be compared to fluoxetine in this trial. Durability of treatment will be monitored over a 1-year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of social phobia

Exclusion Criteria:

* Pervasive developmental disorders (PDD)
* Schizophrenia
* Major Depression
* IQ of less than 80
* Medical conditions contraindicating use of fluoxetine

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 139 (Actual)
Dates: Start 2001-04; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Maryland Center for Anxiety Disorders, University of Maryland, College Park, Maryland, United States

REFERENCES:
- [Result] Beidel DC, Turner SM, Sallee FR, Ammerman RT, Crosby LA, Pathak S. SET-C versus fluoxetine in the treatment of childhood social phobia. J Am Acad Child Adolesc Psychiatry. 2007 Dec;46(12):1622-32. doi: 10.1097/chi.0b013e318154bb57. PMID 18030084
- [Derived] De Los Reyes A, Alfano CA, Beidel DC. Are clinicians' assessments of improvements in children's functioning "global"? J Clin Child Adolesc Psychol. 2011;40(2):281-94. doi: 10.1080/15374416.2011.546043. PMID 21391024
- [Derived] De Los Reyes A, Alfano CA, Beidel DC. The relations among measurements of informant discrepancies within a multisite trial of treatments for childhood social phobia. J Abnorm Child Psychol. 2010 Apr;38(3):395-404. doi: 10.1007/s10802-009-9373-6. PMID 20013046